CLINICAL TRIAL: NCT02432118
Title: A Feasibility Study of Radiofrequency Identification (RFID) Localization of Breast Lesions
Brief Title: Radiofrequency-Guided Localization in Patients With Abnormal Breast Tissue Undergoing Lumpectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient resources
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BRS0053; NCI-2015-00630 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 348; BRS0053 (Other: Stanford University Hospitals and Clinics); P30CA124435 (NIH)
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental; Radio Frequency Identification Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (radiofrequency-guided localization) (Experimental): Patients undergo radiofrequency-guided localization comprising RFID tag placement before lumpectomy and interactive detection of tag using RFID reader during lumpectomy.
  Interventions: Procedure: Lumpectomy; Other: Questionnaire Administration; Procedure: Radiofrequency-Guided Localization

INTERVENTIONS:
Procedure: Lumpectomy — Undergo lumpectomy
  Other Names: Lumpectomy of Breast; partial mastectomy
Other: Questionnaire Administration — Ancillary studies
Procedure: Radiofrequency-Guided Localization — Undergo radiofrequency-guided localization

SUMMARY:
This pilot clinical trial studies the use of the radiofrequency-guided localization in patients with abnormal breast tissue undergoing lumpectomy (a type of breast-sparing surgery). The radiofrequency identification localization system consists of an implantable radiofrequency identification tag and a hand-held radiofrequency reader to mark abnormal breast tissue before surgery and later surgically retrieve them. Radiofrequency-guided localization may make it easier to find and remove abnormal breast tissue during lumpectomy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain human clinical data in order to demonstrate that the Radiofrequency Identification (RFID) Localization System performs as intended as a localization device for marking and retrieving a surgical target in the breast.

SECONDARY OBJECTIVES:

I. To solicit feedback from the radiologists and surgeons regarding the process and use of the RFID system.

OUTLINE:

Patients undergo radiofrequency-guided localization comprising RFID tag placement before lumpectomy and interactive detection of tag using RFID reader during lumpectomy.

ELIGIBILITY:
Inclusion Criteria:

* Have had stereotactic or ultrasound-guided biopsy with marker placement
* Have a lesion or biopsy marker that is visible under ultrasound
* Have a surgical target =< 6 cm from the skin when lying supine
* Have a discreet surgical target
* Have a lesion in which the center/focal area is defined
* Have the ability to understand and the willingness to sign a written informed consent document
* Eastern Cooperative Oncology Group (ECOG)/Karnofsky performance status will not be used as an inclusion criterion
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Require more than one localization needle for localization of the surgical target (bracket localization)
* Have undergone previous open surgical biopsy, lumpectomy, or mastectomy in the operative breast
* Have a prosthesis/implant in the operative breast
* Have a cardiac pacemaker or defibrillator device
* Be contraindicated for surgery
* Be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Localization success, defined as the surgical target visualized in the removed specimen AND the RFID tag removed from the patient's breast | At time of surgery
  Will be summarized using descriptive statistics, including total numbers, percentages, means, and proportions.

SECONDARY OUTCOMES:
Feedback solicited from the radiologist and surgeon | Up to 12 months after lumpectomy
  Feedback solicited from the radiologist and surgeon will be summarized using qualitative methods. Each questionnaire will be reviewed for both positive and negative responses and summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Jafi Lipson, Principal Investigator — Stanford University Hospitals and Clinics